CLINICAL TRIAL: NCT02639689
Title: Evaluation of the Increase of the Driving Speed After the Apparatus by Walkaide® Medical Device in Deficits Levator Foot of Central Origin.
Brief Title: Evaluation of the Increase of the Driving Speed With Walkaide® Medical Device
Acronym: WALKAIDE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU PROMOTEUR 2013/12
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Foot Sensory Deficit
Keywords: Deficits of foot relievers of central origin; Walkaide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WALKAIDE (Experimental): A clinical evaluation will be conducted at T0 with achievement of the following tests without orthosis and with the usual orthosis if applicable: he will be made a stimulation test of common peroneal nerve and settings Walkaide® device.
  Subjects will be reconvened at T1, one to four weeks after the initial assessment to ensure the stability of walking speed. We will perform the following tests without orthosis and with the usual orthosis if applicable. The final evaluation (T2) will be 28 days after the start of the port of the device.
  Interventions: Device: WALKAIDE

INTERVENTIONS:
Device: WALKAIDE — A clinical evaluation will be conducted at T0 with achievement of the following tests without orthosis and with the usual orthosis if applicable: he will be made a stimulation test of common peroneal nerve and settings Walkaide® device.
  Subjects will be reconvened at T1, one to four weeks after the initial assessment to ensure the stability of walking speed. We will perform the following tests without orthosis and with the usual orthosis if applicable. The final evaluation (T2) will be 28 days after the start of the port of the device.

SUMMARY:
Evaluation of the increase of the driving speed after apparatus by Walkaide® medical device in deficits levator foot of central origin.

DETAILED DESCRIPTION:
Evaluation of the increase of the driving speed after apparatus by Walkaide® medical device in deficits levator foot of central origin.

The main objective is the study of changes in walking speed on the 6-minute walk test between the initial walk without orthotic and walking with orthotic Walkaide® medical devie after one month of training.

This is a prospective multicenter study, without control group, qualified as a biomedical research.

ELIGIBILITY:
Inclusion Criteria:

* Passive ankle dorsiflexion of at least 0 ° (strained knee)
* No injection of botulinum toxin in the lower limbs for at months 3 months
* No surgery for at least three months
* Walk 10 meters in less than 60 seconds, without human help, with or without technical assistance
* Score the Functional Ambulation Classification (FAC) ≥ 3
* Ashworth Score ≤ 2 sural triceps
* Written consent signed

Exclusion Criteria:

* Presence of severe cognitive impairment that does not allow the use of the device independently
* History of debilitating disease associated general
* Local embarrassing skin disorder laying the electrodes
* Pacemaker
* Unstable Epilepsy
* Pregnancy and lactation
* Participation Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change in walking speed | One month
  The main objective is the study of changes in walking speed on the 6-minute walk test between the initial walk without orthotics and walking with Walkaide® functionnal electric stimulation orthosis after one month of training.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Richard, md-PHD, Principal Investigator — University Hospital, Angers
Locations (1):
- Les Capucins, Angers, Pays de la Loire Region, France

REFERENCES:
- [Result] Stein RB, Everaert DG, Thompson AK, Chong SL, Whittaker M, Robertson J, Kuether G. Long-term therapeutic and orthotic effects of a foot drop stimulator on walking performance in progressive and nonprogressive neurological disorders. Neurorehabil Neural Repair. 2010 Feb;24(2):152-67. doi: 10.1177/1545968309347681. Epub 2009 Oct 21. PMID 19846759
- [Result] Detrembleur C, Dierick F, Stoquart G, Chantraine F, Lejeune T. Energy cost, mechanical work, and efficiency of hemiparetic walking. Gait Posture. 2003 Oct;18(2):47-55. doi: 10.1016/s0966-6362(02)00193-5. PMID 14654207
- [Result] Kottink AI, Oostendorp LJ, Buurke JH, Nene AV, Hermens HJ, IJzerman MJ. The orthotic effect of functional electrical stimulation on the improvement of walking in stroke patients with a dropped foot: a systematic review. Artif Organs. 2004 Jun;28(6):577-86. doi: 10.1111/j.1525-1594.2004.07310.x. PMID 15153151
- [Result] Everaert DG, Thompson AK, Chong SL, Stein RB. Does functional electrical stimulation for foot drop strengthen corticospinal connections? Neurorehabil Neural Repair. 2010 Feb;24(2):168-77. doi: 10.1177/1545968309349939. Epub 2009 Oct 27. PMID 19861590
- [Result] Sabut SK, Lenka PK, Kumar R, Mahadevappa M. Effect of functional electrical stimulation on the effort and walking speed, surface electromyography activity, and metabolic responses in stroke subjects. J Electromyogr Kinesiol. 2010 Dec;20(6):1170-7. doi: 10.1016/j.jelekin.2010.07.003. Epub 2010 Aug 6. PMID 20692180